CLINICAL TRIAL: NCT05570565
Title: Ultrasound Guided Bilateral Erector Spinae Plane Block Versus Preincisional Local Field Block for Perioperative Analgesia in Lumbar Spine Surgeries; Randomized Controlled Study
Brief Title: Erector Spinae Block Versus Local Field Block in Lumbar Spine Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd elmoneim Adel Abd elmoneim, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-40-2022
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; Erector spinae plane block; lumbar spine surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane group (Experimental): The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of L3. a curvilinear ultrasound transducer will be placed sagittal 3 cm lateral to L3 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 20 mL of local anesthestic mixture of 0.25% bupivacaine and 1%lidocaine adrenaline (1;200000) will be injected. The procedure will be repeated following the same steps on the other side.
  The surgical intervention will be then allowed 20 minutes after finishing the block procedure
  Interventions: Procedure: Erector spinae plane block
- local field block (Active Comparator): For the preincisional local field block, a 23-gauge needle is used to infiltrate 20mL of local anesthestic mixture of 0.25% bupivacaine and 1%lidocaine adrenaline (1;200000) will be injected in the subcutaneous space and in the paravertebral muscles on each side of the spinous processes of the presumed surgical approach.
  Interventions: Procedure: local field block

INTERVENTIONS:
Procedure: Erector spinae plane block — ultrasound guided injection of local anesthestics drugs (mixture of lidocaine and bupivacaine) in the Erector spinae plane which lies between the Erector spinae muscle and lumbar transverse process
  Arms: Erector spinae plane group
Procedure: local field block — infiltration of local anesthestic drugs( mixture of lidocaine and bupivacaine) in the surgical field before surgical incision
  Arms: local field block

SUMMARY:
Major lumbar spine surgeries are associated with significant postoperative pain that may last for days,So In this study, we intend to evaluate if preventive analgesia with a single injection dose of ultrasound guided bilateral erector spinae is a safe and better method of peri-operative analgesia for lumbar spine surgeries than preincisional local field block.

DETAILED DESCRIPTION:
Patients scheduled for lumbar spine surgery will be recruited and a written informed consent will be obtained from patients.

All patients will be assessed clinically and investigated for exclusion of any of the above mentioned contraindications. Laboratory work needed will be: Complete blood count (CBC); prothrombin time and concentration (PT& PC); partial thromboplastin time (PTT); bleeding time (BT); clotting time (CT) , liver function tests and kidney function tests .

● Operating Room preparation & Equipment: The ultrasound used will be curvilinear high-frequency ultrasound transducer (Siemens acuson x300 3-5 MHz ultrasound)

• Methods: General anaesthesia will be induced. 1.5 μg/kg fentanyl based on lean body weight with maximum dose of 200 μg and 2 mg/kg propofol will be given based on total body weight. Tracheal intubation will be facilitated with 0.5 mg/kg atracurium based on ideal body weight.

Volume controlled ventilation will be adjusted to maintain normocapnia . Anesthesia will be maintained by using 1.5% isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes.

Patients will be placed in the prone position on a Relton Hall frame or padded bolsters.

* In group (A): local field block For the preincisional local field block, a 23-gauge needle is used to infiltrate 20mL of local anesthestic mixture of 0.25% bupivacaine and 1%lidocaine adrenaline (1;200000) will be injected in the subcutaneous space and in the paravertebral muscles on each side of the spinous processes of the presumed surgical approach.
* In group (B): Bilateral Ultrasound guided Erector spinae group. The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of L3. a curvilinear high-frequency ultrasound transducer will be placed sagittal 3 cm lateral to L3 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 20 mL of local anesthestic mixture of 0.25% bupivacaine and 1%lidocaine adrenaline (1;200000) will be injected. The procedure will be repeated following the same steps on the other side.

The surgical intervention will be then allowed 20 minutes after finishing the block procedure.

All participants will be given 1 gram of intravenous paracetamol with maximum dose of 4 gm every 24 hour, together with 4 mg ondansetron 10 min prior to the end of surgery for postoperative nausea and vomiting prophylaxis.

Failed block (increase in HR and mean arterial blood pressure (MABP)>20% from base line with skin incision) will be treated by 0.5 ug/kg of fentanyl as top-up doses and increasing isoflurane concentration in case of inadequate response to fentanyl.

After skin closure , the patient will be turned to supine position,then inhalational anesthesia will be discontinued and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered intravenous after return of patient's spontaneous breathing .the patient will be extubated awake, Patients will then be transferred to post anesthesia care unit (PACU) for 60 min to complete recovery and monitoring.

* At any time hypotension (defined as a decrease in mean arterial pressure (MAP) >25% from baseline value or systolic arterial pressure (SAP <100 mmHg)) will be treated with 5 mg IV bolus ephedrine and repeated every 3 minutes until the hypotension resolved. Bradycardia (HR <50 beats per minute) will be treated with atropine 0.5 mg IV.
* Rescue analgesia :

Intra operative:

0.5ug /kg of fentanyl as top-up doses at any time if blood pressure and heart rate increased by more than 20% from baseline reading .

Post-operative :

In the PACU ; VAS will be assessed 15 minutes after extubation and if the score is exceeding 4/10 , rescue analgesia in the form of Nalbuphine 0.1mg/kg will be given .another dose of Nalbuphine 0.1mg/kg can be given in the PACU if the score still more than 4 after 30 minutes of the 1st dose.

After discharging from the PACU; the analgesic plan will be intravenous paracetamol 1gm every 8hours and ketorolac 0.5mg/kg/6hours as a standard regimen , Nalbuphine 0.1mg/kg will be given as rescue analgesia on demand or at any time if VAS score exceeding 4(maximum 20mg per dose and 160mg in 24 hours)

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years old.
* Patients undergoing Lumbar spine surgery (L1-L5).
* American society of anesthesiologists classification (ASA) I and II.
* BMI < 35
* Duration of surgery less than 3 hours

Exclusion Criteria:

* Patient's refusal.
* Bleeding disorders (platelets count < 150,000; INR >1.5; PC< 60%) and coagulopathies.
* Skin lesion, wounds or infection at the injection site.
* Known allergy to local anesthetic drugs.
* Chronic opioid users.
* Patients with pre-operative opioid consumption.
* Patients on long term therapy of Corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
duration of postoperative analgesia | 24 hours
  Time to first analgesic request

SECONDARY OUTCOMES:
cumulative 24 hour opioid consumption | 24 hours
  the amount of Nalbuphine consumed by the patient in the first 24 hours postoperative
pain assessment using VAS score at 15minutes, 30 minutes,1,2,4,8,12,24 hours postoperative | 24 hours
  The visual analog scale(VAS) score is a validated,subjective measure for acute and chronic pain, scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and"worst pain".
presence of any complications | evey 10 minutes intraoperative till end of surgery (up to 2 hours)
  bradycardia,hypotension, arrythmia
patient satisfaction with anesthesia | 24 hours
  11 point score , where 0=unsatisfied and 10=most satisfied
surgeon satisfaction for surgical field accessibility | 2 hours
  likert 5 point scale, where 1=very unsatisfied and 5=vry satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Abdelmoneim A Abdelmoneim, lecturer, Principal Investigator — Anesthesia department , cairo university
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No